CLINICAL TRIAL: NCT00005357
Title: Pulmonary Hypertension--Mechanisms and Family Registry
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4243; R01HL048164 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Lung Diseases; Hypertension, Pulmonary
MeSH Terms: conditions — Lung Diseases; Hypertension, Pulmonary

SUMMARY:
To establish a registry of primary pulmonary hypertension (PPH), a lethal disease which causes progressive obstruction of small pulmonary arteries and to investigate basic mechanisms of the disease.

DETAILED DESCRIPTION:
BACKGROUND:

Primary pulmonary hypertension (PPH) is a serious disease of unknown cause in which small arteries in the lungs become obstructed. Mean survival is less than three years, and women develop PPH twice as commonly as men. It is familial (FPPH) in about 6 percent of cases. The National FPPH Registry was established in 1994 to collect and analyze family history and clinical data from PPH families to better characterize the disease phenotype as well as to identify the underlying genetic etiology. Through the collection of 72 families, FPPH has been shown to be inherited as an autosomal dominant disorder, with incomplete penetrance and genetic anticipation. Micro-satellite marker studies in six families have identified linkage to chromosome 2q31 without evidence of genetic heterogeneity.

DESIGN NARRATIVE:

The study established a national registry of familial PPH (FPPH). The primary goal of the family registry was to establish and expand the database of FPPH pedigrees to definitively establish the mode of inheritance of FPPH, which initial segregation analysis suggested was autosomal dominant. The FPPH family registry provided the framework for the linkage analysis of the molecular search for basic mechanisms of PPH. The investigators developed a tissue bank for specimens (DNA and transformed lymphocytes) from families and patients with pulmonary hypertension, both for their investigations and as a national resource for other interested investigators. Their search used three different approaches to investigate for a FPPH gene locus. First, they performed karyotyping and high resolution chromosome studies to search for a chromosomal translocation, interstitial deletion, or inversion, the finding of which would implicate a specific gene locus. Second, they pursued the proposed association of human leukocyte antigen (HLA) tissue type with familial PPH in a parallel attempt to identify a related locus about which to perform an intensified molecular search, using regional mapping studies of closely linked markers. Finally, they performed linkage analysis in selected PPH families which had the most informative inheritance patterns, using polymerase chain reaction (PCR) based microsatellite markers for selected candidate genes, including those for transforming growth factor beta, endothelin, beta globin, and HLA. An additional promising approach included a search for linkage of FPPH to genes with GC-rich trinucleotide repeats, as had been successful for other diseases with genetic anticipation, including Fragile X syndrome, myotonic dystrophy, and Huntington's disease.

The study was renewed in 1999 through 2003 to expand the registry in order to obtain enough PPH families to localize and clone the PPH gene, and support the DNA bank for these and further studies. Other goals included prospective and biochemical mediator studies of obligate gene carriers, who did not have clinically evident PPH. This aim determined which mediators first became abnormal during developing PPH, and defined the natural history of pre-symptomatic diseases. In addition, the registry broadened its scope to include sporadic PPH patients, including those who had used appetite suppressant medications, who were screened for gene mutations.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1994-04; Primary Completion 1999-03 (Actual); Study Completion 1999-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Loyd — Vanderbilt University

REFERENCES:
- [Background] Loyd JE, Slovis B, Phillips JA 3rd, Butler MG, Foroud TM, Conneally PM, Newman JH. The presence of genetic anticipation suggests that the molecular basis of familial primary pulmonary hypertension may be trinucleotide repeat expansion. Chest. 1997 Jun;111(6 Suppl):82S-83S. doi: 10.1378/chest.111.6_supplement.82s. No abstract available. PMID 9184540
- [Background] Nichols WC, Koller DL, Slovis B, Foroud T, Terry VH, Arnold ND, Siemieniak DR, Wheeler L, Phillips JA 3rd, Newman JH, Conneally PM, Ginsburg D, Loyd JE. Localization of the gene for familial primary pulmonary hypertension to chromosome 2q31-32. Nat Genet. 1997 Mar;15(3):277-80. doi: 10.1038/ng0397-277. PMID 9054941
- [Background] Robbins IM, Christman BW, Newman JH, Matlock R, Loyd JE. A survey of diagnostic practices and the use of epoprostenol in patients with primary pulmonary hypertension. Chest. 1998 Nov;114(5):1269-75. doi: 10.1378/chest.114.5.1269. PMID 9824000
- [Background] Chazova I, Robbins I, Loyd J, Newman J, Tapson V, Zhdaov V, Meyrick B. Venous and arterial changes in pulmonary veno-occlusive disease, mitral stenosis and fibrosing mediastinitis. Eur Respir J. 2000 Jan;15(1):116-22. doi: 10.1183/09031936.00.15111600. PMID 10678631
- [Background] Machado RD, Pauciulo MW, Thomson JR, Lane KB, Morgan NV, Wheeler L, Phillips JA 3rd, Newman J, Williams D, Galie N, Manes A, McNeil K, Yacoub M, Mikhail G, Rogers P, Corris P, Humbert M, Donnai D, Martensson G, Tranebjaerg L, Loyd JE, Trembath RC, Nichols WC. BMPR2 haploinsufficiency as the inherited molecular mechanism for primary pulmonary hypertension. Am J Hum Genet. 2001 Jan;68(1):92-102. doi: 10.1086/316947. Epub 2000 Dec 12. PMID 11115378
- [Background] Thomson JR, Machado RD, Pauciulo MW, Morgan NV, Humbert M, Elliott GC, Ward K, Yacoub M, Mikhail G, Rogers P, Newman J, Wheeler L, Higenbottam T, Gibbs JS, Egan J, Crozier A, Peacock A, Allcock R, Corris P, Loyd JE, Trembath RC, Nichols WC. Sporadic primary pulmonary hypertension is associated with germline mutations of the gene encoding BMPR-II, a receptor member of the TGF-beta family. J Med Genet. 2000 Oct;37(10):741-5. doi: 10.1136/jmg.37.10.741. PMID 11015450
- [Background] International PPH Consortium; Lane KB, Machado RD, Pauciulo MW, Thomson JR, Phillips JA 3rd, Loyd JE, Nichols WC, Trembath RC. Heterozygous germline mutations in BMPR2, encoding a TGF-beta receptor, cause familial primary pulmonary hypertension. Nat Genet. 2000 Sep;26(1):81-4. doi: 10.1038/79226. PMID 10973254
- [Background] Doyle TP, Loyd JE, Robbins IM. Percutaneous pulmonary artery and vein stenting: a novel treatment for mediastinal fibrosis. Am J Respir Crit Care Med. 2001 Aug 15;164(4):657-60. doi: 10.1164/ajrccm.164.4.2012132. PMID 11520733
- [Background] Trembath RC, Thomson JR, Machado RD, Morgan NV, Atkinson C, Winship I, Simonneau G, Galie N, Loyd JE, Humbert M, Nichols WC, Morrell NW, Berg J, Manes A, McGaughran J, Pauciulo M, Wheeler L. Clinical and molecular genetic features of pulmonary hypertension in patients with hereditary hemorrhagic telangiectasia. N Engl J Med. 2001 Aug 2;345(5):325-34. doi: 10.1056/NEJM200108023450503. PMID 11484689
- [Background] Holcomb BW, Loyd JE, Byrd BF 3rd, Wilsdorf TT, Casey-Cato T, Mason WR, Robbins IM. Iatrogenic paradoxical air embolism in pulmonary hypertension. Chest. 2001 May;119(5):1602-5. doi: 10.1378/chest.119.5.1602. PMID 11348976
- [Background] Province MA, Rao DC. General purpose model and a computer program for combined segregation and path analysis (SEGPATH): automatically creating computer programs from symbolic language model specifications. Genet Epidemiol. 1995;12(2):203-19. doi: 10.1002/gepi.1370120208. PMID 7607419
- [Background] Loyd JE. Parker B. Francis Lecture. Genetics and gene expression in pulmonary hypertension. Chest. 2002 Mar;121(3 Suppl):46S-50S. doi: 10.1378/chest.121.3_suppl.46s. No abstract available. PMID 11893683
- [Background] Runo JR, Loyd JE. Primary pulmonary hypertension. Lancet. 2003 May 3;361(9368):1533-44. doi: 10.1016/S0140-6736(03)13167-4. PMID 12737878
- [Background] Loyd JE. Genetics and pulmonary hypertension. Chest. 2002 Dec;122(6 Suppl):284S-286S. doi: 10.1378/chest.122.6_suppl.284s. PMID 12475800
- [Background] Runo JR, Vnencak-Jones CL, Prince M, Loyd JE, Wheeler L, Robbins IM, Lane KB, Newman JH, Johnson J, Nichols WC, Phillips JA 3rd. Pulmonary veno-occlusive disease caused by an inherited mutation in bone morphogenetic protein receptor II. Am J Respir Crit Care Med. 2003 Mar 15;167(6):889-94. doi: 10.1164/rccm.200208-861OC. Epub 2002 Nov 21. PMID 12446270
- [Background] Kuhn KP, Byrne DW, Arbogast PG, Doyle TP, Loyd JE, Robbins IM. Outcome in 91 consecutive patients with pulmonary arterial hypertension receiving epoprostenol. Am J Respir Crit Care Med. 2003 Feb 15;167(4):580-6. doi: 10.1164/rccm.200204-333OC. Epub 2002 Nov 21. PMID 12446266
- [Background] Newman JH, Wheeler L, Lane KB, Loyd E, Gaddipati R, Phillips JA 3rd, Loyd JE. Mutation in the gene for bone morphogenetic protein receptor II as a cause of primary pulmonary hypertension in a large kindred. N Engl J Med. 2001 Aug 2;345(5):319-24. doi: 10.1056/NEJM200108023450502. PMID 11484688